CLINICAL TRIAL: NCT02849158
Title: Interest in Studying Fibroblast Before and After Neoadjuvant Chemo-radiotherapy in Patient With Locally Advanced Rectal Adenocarcinoma : Exploratory Study
Brief Title: Fibroblast Before and After Neoadjuvant Chemo-radiotherapy in Patient With Locally Advanced Rectal Adenocarcinoma
Acronym: FibroRect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2015-12
Record Dates: First submitted 2016-07-13; First posted 2016-07-29 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Rectum Adenocarcinoma
Keywords: Rectoscopy; Proctectomy; Fibroblasts
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy (Experimental): Patients will have new biopsy before starting RT-CT and samples will be taken on rectum surgery at the level of the tumor and away from the rectum.
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Rectoscopy with biopsy

SUMMARY:
Single center interventional study to explore activity of fibroblasts in the tumor and away in the healthy rectal tissue.

DETAILED DESCRIPTION:
Patients included in the trial will have new biopsy performed before starting the Radiation Therapy and Chemotherapy (RT-CT). These biopsies will study the activity of fibroblasts in the tumor and away in the healthy rectal tissue. Within 8 to 10 weeks after the end of RT-CT, patients will have cancer surgery by proctectomy (with complete removal of the meso-rectum). On the resection specimen, new samples will be taken at the level of the tumor and away from the rectum.This study is single center interventional exploratory .

ELIGIBILITY:
Inclusion Criteria:

1. Middle rectum adenocarcinoma Tumor(T)x Node (N)+ or T3 /T4 N0 or N+
2. Classification done on pelvic Magnetic Resonance Imaging (MRI) and rectal ultrasonography
3. Age ≥ 18
4. No contraindication to treatment with capecitabine
5. Able to receive radiotherapy 50 Grays in 5 weeks
6. No contraindication for surgery after chemoradiotherapy which will be 8 to 10 weeks after completion of chemoradiotherapy
7. Patient or legal representative provided with information and signature of informed consent

Exclusion Criteria:

1. High rectum adenocarcinoma
2. Contraindication to rectal biopsy: including anti-coagulants or anti-platelet agents (vitamin K antagonists, clopidogrel, aspirin > 160 grams) that cannot be interrupted
3. Pregnant woman or breastfeeding
4. Persons deprived of their liberty, or under guardianship
5. Impossibility of undergoing the trial's medical follow-up for geographical, social or psychological reasons.
6. Patient already included in another therapeutic trial with an experimental medication during the realization of protocol biopsies and surgery
7. Patient not covered by health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Proteomic level evaluation in intra-tumor fibroblast | 3 years
  Proteomic level is assessed before and after radiochemotherapy using SILAC technic (Stable Isotope Labeling by Amino acids in Cell culture)

SECONDARY OUTCOMES:
Study of fibroblast impact on colorectal tumor cells (in vitro) | 3 years
  In vitro analysis including tumor cells characteristics: proliferation, invasive potential, stem cells phenotype).

OTHER OUTCOMES:
Metastatic spread evaluation | 3 years
  On a mouse model of orthotopic rectal cancer, assessment of the potential and metastatic tumor growth
Outcomes 1 to 3 correlation with histological response after RT-CT | 3 years
  Histological response after RT-CT assessed according to the tumor regression grading - Dworak 1997
Disease-free survival | 5 years
  Disease-free Survival assessment

CONTACTS AND LOCATIONS:
Overall Officials: Pascale MARIANI, LDD, Principal Investigator — Institut Curie
Locations (3):
- France (3):
  - INSTITUT CURIE - Site Paris, Paris
  - Institut Curie, Paris, Île-de-France Region
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accordance with Institut Curie policies.
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).